CLINICAL TRIAL: NCT00235287
Title: Pulse Wave Velocity, Pulse Wave Morphology and Blocking of the Reninangiotensin System in Patients With Chronic Kidney Disease: An Interventional and Methodological Study
Brief Title: Pulse Wave Velocity, Pulse Wave Morphology and Blocking of the Reninangiotensin System in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Marie Frimodt-Møller, MD, Dept. of Nephrology, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAS-block study
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Kidney Failure, Chronic; Cardiovascular Diseases
Keywords: Angiotensin-Converting Enzyme Inhibitors; type 1 angiotensin receptor antagonists; blood pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — candesartan; Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A,AIIA (Active Comparator): 24 weeks of treatment with Candesartan, where Enalapril is added in the last 8 weeks.
  Interventions: Drug: Candesartan and enalapril
- A, ACE-I (Active Comparator): 24 weeks of treatment with Enalapril, where Candesartan is added in the last 8 weeks.
  Interventions: Drug: candesartan and enalapril
- C, AIIA (Active Comparator): 8 weeks of treatment with Candesartan, followed by 8 weeks of treatment with Enalapril. The treatment in the last 8 out of the 24 weeks is a combination of Candesartan and Enalapril.
  Interventions: Drug: candesartan and enalapril
- C, ACE (Active Comparator): 8 weeks of treatment with Enalapril in incremental doses (5,10,20 mg) , followed by 8 weeks of treatment with Candesartan in incremental doses (4,8,16 mg) . The treatment in the last 8 out of the 24 weeks is a combination of Candesartan 16 mg and Enalapril in incremental doses (5,10,20 mg)
  Interventions: Drug: candesartan and enalapril

INTERVENTIONS:
Drug: Candesartan and enalapril — 24 weeks of treatment with Candesartan in incremental doses (4,8,16 mg), where Enalapril is added in incremental doses (5,10 and 20 mg)the last 8 weeks.
  Arms: A,AIIA
Drug: candesartan and enalapril — 24 weeks of treatment with Enalapril in incremental doses (5, 10, 20 mg), where Candesartan is added in incremental doses (4,8,16 mg) in the last 8 weeks.
  Arms: A, ACE-I
Drug: candesartan and enalapril — 8 weeks of treatment with Candesartan in incremental doses (4,8,16 mg), followed by 8 weeks of treatment with Enalapril in incremental doses (/5,10,20 mg). The treatment in the last 8 out of the 24 weeks is a combination of Candesartan in incremental doses (4,8,16 mg) and Enalapril 20 mg.
  Arms: C, AIIA
Drug: candesartan and enalapril — 8 weeks of treatment with Enalapril in incremental doses (5,10,20 mg), followed by 8 weeks of treatment with Candesartan (4,8,16 mg). The treatment in the last 8 out of the 24 weeks is a combination of Candesartan 16 mg and Enalapril in incremental doses (5,10,20 mg)
  Arms: C, ACE

SUMMARY:
The purpose of this study is to determine whether a combination therapy with angiotensin-converting enzyme (ACE)-inhibitors and angiotensin receptor blockers reduces the arterial stiffness assessed by applantiontonometry more than a single treatment in kidney patients.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine: 150-350 micromol/L
* Blood pressure > 110 systolic
* Negative pregnancy test for fertile women
* Written and oral informed consent from the patient

Exclusion Criteria:

* Treatment with both ACE-inhibitors (ACE-I) and angiotensin receptor blockers
* Pregnancy or breastfeeding
* Treatment with immunosuppressive medication, steroids or non-steroidal anti-inflammatory drugs (NSAIDs)
* Serious chronic heart failure (New York Heart Association [NYHA] III-IV)
* Chronic liver disease
* Suspicion or verified kidney artery stenosis
* Cardiac arrhythmia and/or implanted pacemaker
* Myocardial infarction or cerebrovascular incidence within the last 3 months
* Allergy towards ACE-I or angiotensin receptor blockers
* Amputation of a whole extremity or the crural or femoral part of the leg
* Dementia or a psychological condition that makes understanding of the examination conditions impossible
* Dialysis or renal transplantation
* Treatment with aldosterone antagonists
* Hyperkalemia > 5.5 mmol/l
* Another serious chronic non-renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
pulse wave velocity (aortic and brachial) | 0, 8, 16 and 24 weeks after start of intervention

SECONDARY OUTCOMES:
augmentation index | 0, 8, 16 and 24 weeks after start of intervention
blood pressure (brachial and aortic) | 0, 8, 16 and 24 weeks after start of intervention
buckbergs index | 0, 8, 16 and 24 weeks after start of interven
time to reflection | 0, 8, 16 and 24 weeks after start of interven
pulse pressure | 0, 8, 16 and 24 weeks after start of interven
change in glomerular filtration rate (GFR) | 0, 8, 16 and 24 weeks after start of interven
blood parameters | at start of intervention and after each 2.5 - 3.week in the study period

CONTACTS AND LOCATIONS:
Overall Officials: Marie Frimodt-Møller, MD, Principal Investigator — Dept. of Nephrology, Herlev University Hospital
Locations (1):
- Dept. of Nephrology, Herlev University Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Cooper TE, Teng C, Tunnicliffe DJ, Cashmore BA, Strippoli GF. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers for adults with early (stage 1 to 3) non-diabetic chronic kidney disease. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD007751. doi: 10.1002/14651858.CD007751.pub3. PMID 37466151
- [Derived] Frimodt-Moller M, Kamper AL, Strandgaard S, Kreiner S, Nielsen AH. Beneficial effects on arterial stiffness and pulse-wave reflection of combined enalapril and candesartan in chronic kidney disease--a randomized trial. PLoS One. 2012;7(7):e41757. doi: 10.1371/journal.pone.0041757. Epub 2012 Jul 31. PMID 22860014